CLINICAL TRIAL: NCT03005327
Title: A Phase 2, Open-Label, Multi-Center Trial of Mavorixafor in Patients With WHIM Syndrome
Brief Title: A Dose Determination and Safety Study of X4P-001 (Mavorixafor) in Participants With Warts, Hypogammaglobulinemia, Infections, and Myelokathexis (WHIM) Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-MKKA; 2016-005028-26 (EudraCT Number)
Record Dates: First submitted 2016-12-20; First posted 2016-12-29 (Estimated); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: WHIM Syndrome
MeSH Terms: conditions — WHIM syndrome | interventions — mavorixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- X4P-001 (Experimental): Initial Treatment Phase: Participants will initiate treatment with mavorixafor at 50 milligrams (mg) once daily (QD) orally or a higher dose, with potential escalation based on area under the curve for absolute neutrophil count and absolute leukocyte count (AUCANC/ALC) values to a maximum total daily dose of 400 mg. Participants are expected to receive treatment for 24 weeks in the initial Treatment Period or until development of a treatment-limiting toxicity (TLT).
  Extension Phase: All participants will receive mavorixafor; the dose will not exceed 400 mg. In the Extension Phase, treatment may continue until mavorixafor becomes available via an alternative mechanism (for example, drug is commercially available, an expanded access program, etc.) or until the study is terminated by the sponsor.
  Interventions: Drug: X4P-001

INTERVENTIONS:
Drug: X4P-001 — Mavorixafor will be provided as either 25 mg or 100 mg capsules.
  Other Names: AMD11070

SUMMARY:
This is a Phase 2 study with an initial 24-week Treatment Period and an Extension Phase. The primary objectives of this Phase 2 study are to determine the safety, tolerability, and dose selection of mavorixafor in participants with WHIM syndrome. Participants may continue treatment in an Extension Phase, if regionally applicable, until mavorixafor becomes available via an alternative mechanism (for example, drug is commercially available, an expanded access program, etc.) or until the study is terminated by the Sponsor for any reason.

ELIGIBILITY:
Inclusion Criteria:

Participants with a clinical diagnosis of WHIM syndrome must meet all of the following criteria to be eligible for study participation:

1. Be at least 18 years of age.
2. Has signed the current approved informed consent form.
3. Has a genotype-confirmed mutation of chemokine receptor type 4 (CXCR4) consistent with WHIM syndrome.
4. Agree to use effective contraception.
5. Be willing and able to comply with this protocol.
6. Has confirmed ANC less than or equal to (≤) 400/µL or ALC ≤650/µL or both.

Exclusion Criteria:

Participants with any of the following will be excluded from participation in the study:

1. Has known systemic hypersensitivity to the mavorixafor drug substance or its inactive ingredients.
2. Is pregnant or nursing.
3. Has a known history of a positive serology or viral load for human immunodeficiency virus (HIV) or a known history of acquired immunodeficiency syndrome (AIDS).
4. Has, at Screening, laboratory tests meeting one or more of the following criteria:

   * A positive antibody test for hepatitis C virus (HCV), unless documented to have no detectable viral load on 2 independent samples.
   * A positive test for hepatitis B surface antigen (HBsAg).
5. Has any medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the participant, or may preclude the participant's successful completion of the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Washington Medical Center, Seattle, Washington, United States
- St. Vincent's Hospital, Fitzroy, Victoria, Australia

REFERENCES:
- [Derived] Dale DC, Firkin F, Bolyard AA, Kelley M, Makaryan V, Gorelick KJ, Ebrahim T, Garg V, Tang W, Jiang H, Skerlj R, Beaussant Cohen S. Results of a phase 2 trial of an oral CXCR4 antagonist, mavorixafor, for treatment of WHIM syndrome. Blood. 2020 Dec 24;136(26):2994-3003. doi: 10.1182/blood.2020007197. PMID 32870250

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each participant was treated at doses that were increased up to a maximum total daily dose of 400 milligrams (mg) based on their individual area under the curve for absolute neutrophil count and absolute leukocyte count (AUCANC/ALC) values.
Groups:
- X4P-001 50 to up to 400 mg/kg: Participants received X4P-001 (mavorixafor) orally once daily (QD) at doses between 50 mg and 400 mg for the Initial Treatment Period (24 weeks) and could continue participation in the open-label Extension Phase until experiencing a treatment-limiting toxicity (TLT) event, X4P-001 was available commercially, or until the study was terminated by the Sponsor.
- X4P-001 100 to up to 400 mg/kg: Participants received X4P-001 (mavorixafor) orally QD at doses between 100 mg and 400 mg for the Initial Treatment Period (24 weeks) and could continue participation in the open-label Extension Phase until experiencing a TLT event, X4P-001 was available commercially, or until the study was terminated by the Sponsor.
- X4P-001 200 to up to 400 mg/kg: Participants received X4P-001 (mavorixafor) orally QD at doses between 200 mg and 400 mg for the Initial Treatment Period (24 weeks) and could continue participation in the open-label Extension Phase until experiencing a TLT event, X4P-001 was available commercially, or until the study was terminated by the Sponsor.
- X4P-001 300 to up to 400 mg/kg: Participants received X4P-001 (mavorixafor) orally QD at doses between 300 mg and 400 mg for the Initial Treatment Period (24 weeks) and could continue participation in the open-label Extension Phase until experiencing a TLT event, X4P-001 was available commercially, or until the study was terminated by the Sponsor.
Period: Initial Treatment Period (24 Weeks)
Arm/Group | X4P-001 50 to up to 400 mg/kg | X4P-001 100 to up to 400 mg/kg | X4P-001 200 to up to 400 mg/kg | X4P-001 300 to up to 400 mg/kg
Started | 2 | 2 | 2 | 2
Received at Least 1 Dose of Study Drug | 2 | 2 | 2 | 2
Completed | 2 | 1 | 1 | 2
Not Completed | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Extension Phase (56 Months)
Arm/Group | X4P-001 50 to up to 400 mg/kg | X4P-001 100 to up to 400 mg/kg | X4P-001 200 to up to 400 mg/kg | X4P-001 300 to up to 400 mg/kg
Started | 2 | 0 (Participant discontinued the study prior to the initiation of extension phase due to unknown reason.) | 1 | 2
Completed | 2 | 0 | 1 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received at least 1 dose of the study medication (mavorixafor). Per prespecified analysis, data were collected for the 'Baseline Characteristics' as a single Arm/Group for any participants who received at least 1 dose of the study drug, regardless of their dose level. Due to the small number of participants per dose, data are reported for the 'Baseline Characteristics' as a single Arm/Group to maintain participant confidentiality.
Groups:
- X4P-001: Participants received X4P-001 (mavorixafor) orally QD at doses between 50 mg and 400 mg for the Initial Treatment Period (24 weeks) and could continue participation in the open-label Extension Phase until experiencing a TLT event, X4P-001 was available commercially, or until the study was terminated by the Sponsor.
Arm/Group | X4P-001
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Value of the Area Under the Plasma Concentration-time Curve for Absolute Neutrophil Count (AUCANC)
Description: AUCANC was collected over a 24-hour period above clinically meaningful thresholds for the mavorixafor-treated participants over 6 months. The absolute neutrophil count (ANC) clinically meaningful threshold was defined as ANC ≥ 600/microliter (μL).
Time Frame: Time 0 (-15 minutes [min] pre-dose), 30, 60, and 90 min (each ± 5 min) and 2, 3, 4, 8, 12, 16, and 24 hours (each ±15 min) at Weeks 5, 13, and 21
Population: Overall Number of Participants Analyzed=number of participants in safety population (all participants who received at least 1 dose of study medication). 'Number analyzed'=number of participants with data above clinically meaningful thresholds at specified timepoints. Participants included in 1 category may be different than participants in other categories. Data for this Outcome Measure were collected by dose level; therefore, participants may have been included in more than 1 arm (dose level).
Measure: Mean (Standard Deviation); unit: cells*hour/μL
Groups:
- X4P-001 50 mg: Participants received X4P-001 50 mg orally QD.
- X4P-001 100 mg: Participants received X4P-001 100 mg orally QD.
- X4P-001 150 mg: Participants received X4P-001 150 mg orally QD.
- X4P-001 200 mg: Participants received X4P-001 200 mg orally QD.
- X4P-001 300 mg: Participants received X4P-001 300 mg orally QD.
- X4P-001 400 mg: Participants received X4P-001 400 mg orally QD.
- X4P-001 300/400 mg: Participants received X4P-001 300 mg or 400 mg orally QD.
Arm/Group | X4P-001 50 mg | X4P-001 100 mg | X4P-001 150 mg | X4P-001 200 mg | X4P-001 300 mg | X4P-001 400 mg | X4P-001 300/400 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 4 | 0 | 4
cells*hour/μL
  Week 5: number analyzed (Participants) | 2 | 2 | 0 | 1 | 2 | 0 | 2
  Week 5 | -12574.63 (156.094) | -6206.75 (4238.280) |  | -6949.58 | 24175.00 (777.817) |  | 24175.00 (777.817)
  Week 13: number analyzed (Participants) | 0 | 2 | 0 | 2 | 1 | 0 | 1
  Week 13 |  | -11291.96 (1509.496) |  | -7575.21 (2701.443) | -2602.50 |  | -2602.50
  Week 21: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0 | 4
  Week 21 |  |  | -8723.00 (2695.962) |  | 58118.02 (112851.505) |  | 58118.02 (112851.505)

2. Primary Outcome: All Visits: Average Per-Participant Value of the AUCANC
Description: AUCANC was collected over a 24-hour period above clinically meaningful thresholds for the mavorixafor-treated participants over 6 months. The ANC clinically meaningful threshold was defined as ANC ≥ 600/μL.
  Data for this outcome measure are reported as an "All Visits" summary based on the mean of AUCs that is, the per-participant average of the AUCANC across the 3 visits where participant was treated with at least 300/400 mg dose. Time frame reported is based on data collection time points.
Time Frame: Time 0 (-15 min pre-dose), 30, 60, and 90 min (each ± 5 min) and 2, 3, 4, 8, 12, 16, and 24 hours (each ±15 min) at Weeks 5, 13, and 21
Population: The Safety Population included all participants who received at least 1 dose of the study medication (mavorixafor). Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: cells*hour/μL
Arm/Group | X4P-001 300/400 mg
Number analyzed (Participants) | 5
cells*hour/μL | 27477.00 (55792.377)

3. Primary Outcome: Mean Value of the Area Under the Plasma Concentration-time Curve for Absolute Lymphocyte Count (AUCALC)
Description: AUCALC was collected over a 24-hour period above clinically meaningful thresholds for the mavorixafor-treated participants over 6 months. The absolute lymphocyte count (ALC) clinically meaningful threshold was defined as ALC ≥ 1000/μL.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cells*hour/μL
Arm/Group | X4P-001 50 mg | X4P-001 100 mg | X4P-001 150 mg | X4P-001 200 mg | X4P-001 300 mg | X4P-001 400 mg | X4P-001 300/400 mg
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 4 | 0 | 4
cells*hour/μL
  Week 5: number analyzed (Participants) | 2 | 2 | 0 | 1 | 2 | 0 | 2
  Week 5 | -5839.54 (6485.407) | 6978.25 (7435.935) |  | 4783.33 | 21837.50 (24236.085) |  | 21837.50 (24236.085)
  Week 13: number analyzed (Participants) | 0 | 2 | 0 | 2 | 1 | 0 | 1
  Week 13 |  | -1006.50 (10546.262) |  | 7023.83 (1603.482) | 2862.50 |  | 2862.50
  Week 21: number analyzed (Participants) | 0 | 0 | 2 | 0 | 4 | 0 | 4
  Week 21 |  |  | -2216.17 (8285.642) |  | 15331.35 (21250.202) |  | 15331.35 (21250.202)

4. Primary Outcome: All Visits: Average Per-Participant Value of the AUCALC
Description: AUCALC was collected over a 24-hour period above clinically meaningful thresholds for the mavorixafor-treated participants over 6 months. The ALC clinically meaningful threshold was defined as ALC ≥ 1000/μL.
  Data for this outcome measure are reported as an "All Visits" summary based on the mean of AUCs that is, the per-participant average of the AUCALC across the 3 visits where participant was treated with at least 300/400 mg dose. Time frame reported is based on data collection time points.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells*hour/μL
Arm/Group | X4P-001 300/400 mg
Number analyzed (Participants) | 5
cells*hour/μL | 14232.17 (16789.700)

5. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence that developed or worsened in severity during the conduct of a clinical study and did not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A TEAE was defined as any AE that began or worsened in severity or frequency on or after the start of study drug through 10 days after the last dose of the study drug. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: From first dose of study drug through 10 days after the last dose of the study drug (Maximum exposure: 1712 days)
Population: The Safety Population included all participants who received at least 1 dose of the study medication (mavorixafor). Data for this Outcome Measure were collected by dose level; therefore, participants may have been included in more than one arm (dose level).
Measure: Count of Participants; unit: Participants
Groups:
- Overall Participants: Participants received X4P-001 (mavorixafor) orally QD at doses between 50 mg and 400 mg for the Initial Treatment Period (24 weeks) and could continue participation in the open-label Extension Phase until experiencing a TLT event, X4P-001 was available commercially, or until the study was terminated by the Sponsor.
Arm/Group | X4P-001 50 mg | X4P-001 100 mg | X4P-001 150 mg | X4P-001 200 mg | X4P-001 300 mg | X4P-001 400 mg | Overall Participants
Number analyzed (Participants) | 2 | 4 | 3 | 4 | 7 | 5 | 8
Participants | 2 | 2 | 2 | 2 | 6 | 3 | 7

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 10 days after the last dose of the study drug (Maximum exposure: 1712 days)
Description: The Safety Population included all participants who received at least 1 dose of the study medication (mavorixafor). All-Cause Mortality and Adverse Event data were collected by dose level; therefore, participants may have been included in more than one arm (dose level).
Arm/Group | X4P-001 50 mg | X4P-001 100 mg | X4P-001 150 mg | X4P-001 200 mg | X4P-001 300 mg | X4P-001 400 mg | Overall Participants
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/4 | 0/7 | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 0/3 | 0/4 | 2/7 | 1/5 | 3/8
Other Adverse Events (participants affected / at risk) | 2/2 | 2/4 | 2/3 | 2/4 | 6/7 | 3/5 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | X4P-001 50 mg (N=2) | X4P-001 100 mg (N=4) | X4P-001 150 mg (N=3) | X4P-001 200 mg (N=4) | X4P-001 300 mg (N=7) | X4P-001 400 mg (N=5) | Overall Participants (N=8)
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | X4P-001 50 mg (N=2) | X4P-001 100 mg (N=4) | X4P-001 150 mg (N=3) | X4P-001 200 mg (N=4) | X4P-001 300 mg (N=7) | X4P-001 400 mg (N=5) | Overall Participants (N=8)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 4
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Genital herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Infected bite (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 2
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 3
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Papilloma viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2 | 3
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 3
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Incision site ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Uterine spasm (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vulva cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/27/NCT03005327/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03005327/SAP_001.pdf